CLINICAL TRIAL: NCT01268124
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HTC-867 Administered Orally to Healthy Japanese Male Subjects
Brief Title: Study Evaluating The Safety and Tolerability of HTC-867 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3253A1-1001-JA
Record Dates: First submitted 2010-01-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: Japanese
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: HTC-867

INTERVENTIONS:
Drug: HTC-867

SUMMARY:
This is a phase 1, randomized (a process that is used to decide whether you will take study drug or a placebo during the study), inpatient study which will assess the safety and tolerability of HTC-867 in healthy male Japanese subjects.

ELIGIBILITY:
Inclusion:

1. Men aged 20 to 45 years inclusive at screening. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after test article administration.
2. Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight ≥45 kg.

   BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's height, in meters, at screening: BMI = Weight (kg)/[Height (m)]2.
3. Healthy as determined by the investigator on the basis of screening evaluations.
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
5. Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

Medical History

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any unstable medical condition.
3. History of seizures.
4. History of cardiac disorders (other than hypertension) including but not limited to valvular disease, congestive heart failure, angina pectoris, myocardial infarction, or arrhythmia.
5. Any significant cardiovascular disease, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
6. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article (eg, resection of liver, kidney, gallbladder, or gastrointestinal tract).
7. Acute disease state (eg, nausea, vomiting, infection, fever, or diarrhea) within 7 days before study day 1).
8. History of drug abuse within 1 year before study day 1.
9. Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements.

   Physical and Laboratory Findings
10. Clinically significant electrocardiogram (ECG) abnormalities.
11. Any clinically important deviation from normal limits in physical examination findings, vital sign measurements, 12-lead ECGs, or clinical laboratory test results.
12. Positive serologic findings for human immunodeficiency virus (HIV) antigen and antibodies, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibodies.
13. Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates, and phencyclidine [PCP]).
14. Troponin T or CK-MB levels above reference range at screening. Allergies and Adverse Drug Reactions
15. History of any clinically important drug allergy (eg, relapsing dermatitis, drug hypersensitivity, drug allergy, hypersensitivity to ingredient in the test articles, angioedema).

    Prohibited Treatments
16. Use of any investigational drug within 90 days before study day 1 or prescription drug within 30 days before study day 1.
17. Tobacco use or the consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or carbonated beverages) or alcoholic beverages within 72 hours before study day 1 until the end of the inpatient confinement period.
18. Consumption of grapefruit or grapefruit-containing products within 72 hours before study day 1 until the end of the inpatient confinement period.
19. Use of any over-the-counter drugs, including herbal supplements (except for the occasional use of vitamins ≤100% of the recommended daily allowance), within 14 days before study day 1 (St. John wort is prohibited within 30 days of study day 1).
20. Donation of blood within 90 days before study day 1. Others
21. Subjects deemed by the investigator to be inappropriate according to the inclusion criteria in the study and according to the screening examination.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety will be measured by vitals signs, labs and electrocardiograms (ECG's). | 7 months

SECONDARY OUTCOMES:
Pharmacokinetics. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer